CLINICAL TRIAL: NCT03500757
Title: Intra-procedural 360-degree Display for Performing Percutaneous Liver Tumor Ablation as an Adjunct to Standard Flat Panel Display
Brief Title: Intra-procedural 360-degree Display for Performing Percutaneous Liver Tumor Ablation
Status: Completed | Type: Observational
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: CASE1218
Record Dates: First submitted 2018-04-10; First posted 2018-04-18 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Percutaneous Tumor Ablation
Keywords: HoloLens; 3D holographic guidance

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- 360-degree Display of solid tumors: Evaluate the feed back of using the HoloLens headset to have a 360 degree visualization of patient tumors during percutaneous liver tumor ablation
  Interventions: Device: HoloLens

INTERVENTIONS:
Device: HoloLens — use the HoloLens to evaluate new 3D holographic guidance and navigation for percutaneous ablation of solid tumors
  Other Names: headset

SUMMARY:
Medical images used to guide treatment of tumor(s) are presently displayed on flat-panel monitors (like screens used with computers). This protocol will evaluate, using a new headset to view the images in true 3D ("360 degrees"), while using standard flat panel monitors as usual (in accordance with standard of care). The headset is combined with a mini-global positioning system (GPS)-like system to help navigate to treat tumor(s). This evaluation is to show that the headset has potential to provide guidance and navigation information that can improve the treatment of tumor(s) with heat.

DETAILED DESCRIPTION:
This protocol will clinically evaluate new 3D holographic guidance and navigation for percutaneous ablation of solid tumors to ultimately overcome limitations of displaying images on 2D flat-panel monitors ("flat screens"). 3D Holographic percutaneous ablation (3D HPA) provides real-time, 360° visualization for guidance and navigation of tracked interventional instruments augmented to the operative site. In this preliminary protocol, 3D HPA will be evaluated as an adjunct to flat-screen display of conventional images used for guidance (ultrasound, fluoroscopy, CT), in accordance with standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Not pregnant
* Willing and able to give informed consent prior to enrollment. This includes media release form.
* Has met all criteria to undergo percutaneous tumor ablation.

Exclusion Criteria:

* Not willing or able to give informed consent
* Patients with pacemakers or automated implantable cardioverter defibrillator (AICDs).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This device evaluation will include patients undergoing percutaneous thermal ablation of solid liver tumors at Cleveland Clinic as clinically indicated in the standard of care.
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2018-04-29 (Actual); Primary Completion 2020-08-17 (Actual); Study Completion 2022-05-16 (Actual)

PRIMARY OUTCOMES:
Standard System Usability Score on a Likert Scale | 1 day
  The surgeons and staff completing the intervention will rate the usability of the system. An average score greater than 3 will indicate acceptability of the 360 degree display.

CONTACTS AND LOCATIONS:
Overall Officials: Charles Martin III, MD, Principal Investigator — Cleveland Clinic, Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic, Case Comprehensive Cancer Center, Cleveland, Ohio, United States